CLINICAL TRIAL: NCT02830308
Title: Evaluation of Adults With Endocrine-Related Conditions
Brief Title: Evaluation of Adults With Endocrine and Metabolic-Related Conditions
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160125; 16-DK-0125
Record Dates: First submitted 2016-07-09; First posted 2016-07-12 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01-14

CONDITIONS: Endocrine Diseases
Keywords: Hormones; Endocrine; Hypercortisolism; Bone; Hypothalamic-Pituitary Dysfunction; Natural History
MeSH Terms: conditions — Endocrine System Diseases; Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with known or suspected endocrine or metabolic dissorde: Adults with known or suspected endocrine or metabolic dissorders

SUMMARY:
Background:

There are many endocrine and metabolic-related conditions. Two well-known disorders include diabetes and thyroid disease. Some of these diseases are caused by a change in genes. Researchers want to identify the genes involved in these disorders. They hope this will help them learn more about these diseases.

Objectives:

To learn more about conditions that affect the hormone-secreting glands (endocrine glands) in adults. To train doctors to diagnose and treat people with endocrine or metabolic conditions.

Eligibility:

Adults age 18 years and older with a known or suspected endocrine disorder.

Relatives ages 18 years and older.

Doctors will review all requests and available medical records to determine final eligibility for the protocol.

Design:

Participants will have a medical history and physical exam.

Most participants will have 1 visit, and may have follow up visits if necessary. They may have tests, surgery, or other procedures to help diagnose or treat their condition. These could include:

* Blood, urine, and saliva tests
* Imaging tests. These may include X-ray, ultrasound, or scans.
* Sleep study
* Medical photographs
* Visits with other specialists at NIH

Participants will provide blood, urine, saliva, or tissue samples. Some of these samples may be stored in the freezer for future studies.

Participants may be asked to participate in genetic testing. They will give a blood or saliva sample for this.

DETAILED DESCRIPTION:
This is an observational protocol designed to collect data from adult subjects with known or suspected endocrine or metabolic disorders.

OBJECTIVE: The overall purpose of endocrine evaluations under this protocol is to increase knowledge of endocrine or metabolic diseases. Adults with known or suspected endocrine or metabolic-related condition(s) may be evaluated under this protocol for:

1. Collection of data for endocrine related conditions (case reports, case series)
2. Collection of data for future research
3. Collection of samples, including leftover samples from clinically indicated tests, for future research (including genomics)

METHODS: Patients will undergo a history and physical exam, anthropometrics, vital signs and endocrine laboratory studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants with known or suspected endocrine disorder age 18 years and older are eligible for this protocol. Protocol investigators will make the actual selection of subjects most appropriate for clinical evaluation.
* Relatives ages 18 years and older may be enrolled if clinically indicated for the diagnosis of a proband.

EXCLUSION CRITERIA:

* Anyone under the age of 18 years old
* Any medical, physical, psychiatric, or social conditions, which, in the opinion of the investigators, would make participation in this protocol not in the best interest of the subject. Subjects who are critically ill, unstable, or with severe organ failure that may affect/limit the endocrine evaluation and place unsustainable demands on Clinical Center or NIDDK resources.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2016-07-09 (Actual); Primary Completion 2029-12-20 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruit a diverse population of adult subjects with a known or suspected endocrine or metabolic disorder in order to provide NIDDK investigators and trainees with hands-on experience related to the diagnosis, management, treatment, and follow-up... | 12/31/2036
  The overall purpose of endocrine evaluations under this protocol is to support our clinical training and research missions.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa F Lightbourne, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified results from clinical trials will be posted on cctrials.gov
Supporting Information: Study Protocol
Time Frame: Not otherwise specified in protocol.
Access Criteria: Only investigators will have access to the data. Publications will not include subject names, nor will they contain personal identifying information. De-identified results from clinical trials will be posted on cctrials.gov

REFERENCES:
- [Derived] Abd-Elmoniem KZ, Edwan JH, Dietsche KB, Villalobos-Perez A, Shams N, Matta J, Baumgarten L, Qaddumi WN, Dixon SA, Chowdhury A, Stagliano M, Mabundo L, Wentzel A, Hadigan C, Gharib AM, Chung ST. Endothelial Dysfunction in Youth-Onset Type 2 Diabetes: A Clinical Translational Study. Circ Res. 2024 Aug 30;135(6):639-650. doi: 10.1161/CIRCRESAHA.124.324272. Epub 2024 Jul 29. PMID 39069898
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-DK-0125.html